CLINICAL TRIAL: NCT02004535
Title: Clinical Study of Cochlear Implants in Adults With Asymmetrical Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201605131; R01DC009010 (NIH)
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Hearing Loss
Keywords: Hearing loss; Asymmetric hearing loss; Cochlear implantation
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear implantation (Experimental): Cochlear implantation of the ear with severe to profound hearing loss
  Interventions: Procedure: Cochlear Implantation

INTERVENTIONS:
Procedure: Cochlear Implantation — The standard surgical procedure for a cochlear implant will be used. The asymmetric participant will receive the cochlear implant in the deaf ear.

SUMMARY:
The objective of this study is to investigate benefits of binaural hearing for non-traditional cochlear implant candidates (with Asymmetric Hearing Loss). Asymmetric candidates are patients with severe to profound hearing loss in one ear and better hearing in the other ear. (One ear is deaf and the other ear has better hearing and in most cases uses a hearing aid.) The investigators hypothesize that cochlear implantation of the poorer ear provides a functional increase in word and sentence understanding in quiet or noise, perceived benefit, localization ability, and other measures of auditory performance relative to use of the better hearing ear alone.

DETAILED DESCRIPTION:
Multichannel cochlear implants have been highly successful in restoring speech understanding in adults and children who have congenital or acquired bilateral profound or severe-to-profound sensorineural (permanent) hearing loss. As implant technology has continued to develop and post-implant performance of patients has improved, the patient selection criteria has broadened to include patients with less severe hearing loss. Further, results from studies where patients received bilateral cochlear implants have demonstrated not only improved performance but the feasibility of integrating signals from both ears.

In contrast to persons with bilateral severe-to-profound hearing loss, persons who have only one ear with profound or severe-to-profound hearing loss and the other ear with substantially less hearing loss have not, to date, been considered cochlear implant candidates. This is because it has been assumed they will do well enough with a conventional hearing aid in the better ear. A problem with this assumption is that even with an appropriately fit better ear hearing aid, many of these hearing-impaired individuals still experience significant difficulties in speech understanding in their everyday listening environments, along with significant communication handicaps that interfere with their employment and quality of life.

Previous studies that have examined the performance of patients who have more symmetrical hearing loss and who wear a cochlear implant on one ear and a power hearing aid on the other ear, have illustrated that the two inputs can be combined and provide binaural hearing benefits. It is hypothesized in this study that patients with an asymmetrical sensorineural hearing loss may also receive significant binaural benefit from having a cochlear implant on the poorer ear along with an appropriately fit hearing aid on the better ear. That is, this study examines whether patients with asymmetrical sensorineural hearing loss can utilize both types of input (acoustic to one ear and electric to the other) effectively, and combine them to receive binaural hearing assistance for improving speech understanding, localization ability, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of surgery
* The poorer ear (implant ear) will have a severe-to-profound hearing loss and meet current cochlear implant candidacy criteria.
* The better ear (contralateral ear) will have hearing levels less than current cochlear implant candidacy criteria and stable/non-fluctuating hearing levels for at least the previous year
* Normal/patent cochlear anatomy
* Fluent in English
* Desire to have more functional binaural hearing and willingness to comply with all of the study requirements

Exclusion Criteria:

* Medical or psychological conditions that contraindicate undergoing surgery
* Additional handicaps that would prevent or restrict participation in the audiological evaluations
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
* Hearing loss of neural or central origin, including auditory neuropathy
* Chronic and severe tinnitus in the ear to be implanted
* Unwillingness or inability to comply with all investigational requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-04; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Sound localization using a 140 degree, horizontal plane loudspeaker arc | Change from Pre-implant baseline localization at 12 months post-implant
  Sound localization using a 140 degree, horizontal plane loudspeaker arc

SECONDARY OUTCOMES:
Speech recognition | Pre-implant and 1, 3, 6, 9, 12, and 24 months post-implant
  Speech recognition will be assessed with word and sentence material for the each ear individually as well as bilaterally (both ears together). Testing will be completed in quiet and in the presence of background noise.
Perceived benefit questionnaire | Pre-implant and 1, 3, 6, 12, and 24 months post-implant
  Speech, Spatial and Qualities of Hearing scale (SSQ; Gatehouse and Noble,2004) will be completed by participants. The SSQ is a 49-item questionnaire that uses a 10-point rating scale (where a 0 rating reflects least ability and 10 reflects greatest ability) to evaluate the effects of hearing loss in terms of disability and function across three domains: Speech Hearing, Spatial Hearing, and Qualities of Hearing.

OTHER OUTCOMES:
Cognitive ability (processing speed, visuospatial working memory, and perceptual effort) | Pre-implant and 12 months post-implant
  processing speed, visuospatial working memory, and perceptual effort

CONTACTS AND LOCATIONS:
Overall Officials: Jill B Firszt, PhD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Firszt JB, Holden LK, Reeder RM, Cowdrey L, King S. Cochlear implantation in adults with asymmetric hearing loss. Ear Hear. 2012 Jul-Aug;33(4):521-33. doi: 10.1097/AUD.0b013e31824b9dfc. PMID 22441359
- [Result] Asymmetric hearing loss. Extended abstracts from the Cochlear Science and Research Seminar. Interlaken, Switzerland. February 10-11, 2011. Audiol Neurootol. 2011;16 Suppl 1:1-26. doi: 10.1159/000327759. No abstract available. PMID 21527825